CLINICAL TRIAL: NCT01109550
Title: Biliary Candidiasis - Evaluation of Risk Factors, Implementation of an Algorithm in Diagnostics and Therapy
Brief Title: Biliary Candidiasis - Optimization of Diagnostics and Therapy
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BILIARY-CANDIDIASIS_2010
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2022-11-28 (Actual); Status verified 2012-12

CONDITIONS: Secondary Cholangitis; Bile Duct Strictures of Unknown Origin
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bile samples, buccal smears, stool samples, blood samples, transpapillary biopsies (bile duct)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with biliary candidiasis: Patients with positive fungal cultures of bile samples.
  Interventions: Procedure: ERCP
- without biliary candidiasis: Patients with negative fungal cultures of bile samples.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — endoscopic retrograde cholangiopancreatography transpapillary biopsies

SUMMARY:
Biliary obstruction and cholangitis are common problems in gastroenterology and need specific therapeutic interventions. Besides a variety of potential causes, infections of the biliary tract with Candida and other fungal species have increasingly been reported in the last few years. Especially interesting is the question, if patients with positive fungal cultures of bile samples should be treated or not and under which circumstances. The primary aim of the present study is to evaluate wether positive fungal cultures of bile samples indicate fungal infection of the biliary tract, rather colonization or simply contamination during endoscopic retrograde cholangiopancreatography (ERCP) procedure.

DETAILED DESCRIPTION:
Background:

Biliary obstruction and cholangitis are common problems in gastroenterology and need specific therapeutic interventions. Besides a variety of potential causes, infections of the biliary tract with Candida and other fungal species have increasingly been reported in the last few years [1-6]. Fungal infections can even lead to common bile duct (CBD) obstruction, as previously reported [7]. Because of the difficulty of gaining bile samples, little is known about the microbial flora of the bile. In a first prospective, observational study, 123 consecutive patients undergoing ERCP for various indications were screened for fungal species [8]. According to this data Candida species may be very frequently be detected in the bile (54/123 patients, 44 % of the cases). As significant risk factors immunosuppression and long-term antibiotic therapy were identified. The main issue in this context is whether positive diagnostic findings represent fungal infection or fungal colonization. Especially interesting is the question, if patients with positive fungal cultures of bile samples should be treated or not and under which circumstances.

Study Aim:

The primary aim of the present study is to evaluate wether positive fungal cultures of bile samples indicate fungal infection of the biliary tract, rather colonization or simply contamination during ERCP procedure. In addition to mycological analysis of bile samples, tissue samples of the common bile duct are collected to confirm fungal invasion.

Study design:

The study is designed as a single-center, non-randomized, observational study. The conducting center is the University Hospital of Muenster, Department of Medicine B, Gastroenterology. The examinations are performed by two experienced gastroenterologists (D. D., H. U.).

Endoscopic Retrograde Cholangiopancreatography (ERCP) procedure:

ERCP is performed using a conventional duodenoscope as described in the literature. To exclude contamination artefacts, smears of the endoscope working channel (elevator) will be taken before and after the examination. Furthermore buccal smears and stool samples will be taken to get an impression of the individual transient flora. Endoscopic transpapillary bile duct biopsy for diagnosing an invasive fungal infection will be performed. Transpapillary biopsies as confirmed by the present literature cause no increased risk for post-interventional bleeding and infection [9-12]. Additionally with routinely taken blood samples (hemoglobin and lipase), candida-antigen-serology and blood-cultures will be gained.

Ethics:

The study protocol conformed to the ethical guidelines of the 1975 Declaration of Helsinki and was a priori approved by the local ethics committee of the University of Muenster.

Statistical methods:

The data will be analyzed using standard statistical methods. As observational study, no power-analysis will reasonable - nevertheless data will be shown with confidence interval. All statistical analyses will be performed in cooperation with the Department of Medical Informatics and Biomathematics.

ELIGIBILITY:
Inclusion Criteria:

* Secondary cholangitis
* Bile duct strictures of unknown origin
* Age ≥ 18 years
* All individuals provide written informed consent before entering the trial

Exclusion Criteria:

* Exclusion criteria and contraindications of the performed procedure
* Ineffective aspiration of bile samples
* Pregnant or breastfeeding patient
* Age < 18 years
* Missing informed consent
* Missing cooperation (language barrier, amblyacousia, psychiatric disease)
* Refusal of participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a hospital of maximum care.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Diagnosis of an invasive fungal infection of the biliary tract | 12 month
  Diagnosis of an invasive fungal infection of the biliary tract

SECONDARY OUTCOMES:
Evaluation of risk factors 2. Implementation of an algorithm in diagnostics and therapy | 12 month
  Risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lenz, M.D., Study Chair — University Hospital of Muenster; Dirk Domagk, M.D., Study Chair — University Hospital of Muenster
Locations (1):
- Unitersity Hospital of Muenster, Department of Medicine B, Münster, Germany

REFERENCES:
- [Background] Banerjee SN, Emori TG, Culver DH, Gaynes RP, Jarvis WR, Horan T, Edwards JR, Tolson J, Henderson T, Martone WJ. Secular trends in nosocomial primary bloodstream infections in the United States, 1980-1989. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):86S-89S. doi: 10.1016/0002-9343(91)90349-3. PMID 1928197
- [Background] Bouche H, Housset C, Dumont JL, Carnot F, Menu Y, Aveline B, Belghiti J, Boboc B, Erlinger S, Berthelot P, et al. AIDS-related cholangitis: diagnostic features and course in 15 patients. J Hepatol. 1993 Jan;17(1):34-9. doi: 10.1016/s0168-8278(05)80518-5. PMID 8445217
- [Background] Domagk D, Fegeler W, Conrad B, Menzel J, Domschke W, Kucharzik T. Biliary tract candidiasis: diagnostic and therapeutic approaches in a case series. Am J Gastroenterol. 2006 Nov;101(11):2530-6. doi: 10.1111/j.1572-0241.2006.00663.x. Epub 2006 Oct 4. PMID 17029620
- [Background] George J, Baillie J. Contemporary Management of Biliary Tract Infections. Curr Infect Dis Rep. 2005 Mar;7(2):108-114. doi: 10.1007/s11908-005-0069-y. PMID 15727737
- [Background] Singh N, Wagener MM, Marino IR, Gayowski T. Trends in invasive fungal infections in liver transplant recipients: correlation with evolution in transplantation practices. Transplantation. 2002 Jan 15;73(1):63-7. doi: 10.1097/00007890-200201150-00011. PMID 11792979
- [Background] Wig JD, Singh K, Chawla YK, Vaiphei K. Cholangitis due to candidiasis of the extra-hepatic biliary tract. HPB Surg. 1998;11(1):51-4. doi: 10.1155/1998/75730. PMID 9830582
- [Background] Domagk D, Bisping G, Poremba C, Fegeler W, Domschke W, Menzel J. Common bile duct obstruction due to candidiasis. Scand J Gastroenterol. 2001 Apr;36(4):444-6. doi: 10.1080/003655201300051397. PMID 11336173
- [Background] Lenz P, Conrad B, Kucharzik T, Hilker E, Fegeler W, Ullerich H, Heinecke A, Domschke W, Domagk D. Prevalence, associations, and trends of biliary-tract candidiasis: a prospective observational study. Gastrointest Endosc. 2009 Sep;70(3):480-7. doi: 10.1016/j.gie.2009.01.038. Epub 2009 Jun 24. PMID 19555935
- [Background] Domagk D, Poremba C, Dietl KH, Senninger N, Heinecke A, Domschke W, Menzel J. Endoscopic transpapillary biopsies and intraductal ultrasonography in the diagnostics of bile duct strictures: a prospective study. Gut. 2002 Aug;51(2):240-4. doi: 10.1136/gut.51.2.240. PMID 12117887
- [Background] Kubota Y, Takaoka M, Tani K, Ogura M, Kin H, Fujimura K, Mizuno T, Inoue K. Endoscopic transpapillary biopsy for diagnosis of patients with pancreaticobiliary ductal strictures. Am J Gastroenterol. 1993 Oct;88(10):1700-4. PMID 8213710
- [Background] Sugiyama M, Atomi Y, Wada N, Kuroda A, Muto T. Endoscopic transpapillary bile duct biopsy without sphincterotomy for diagnosing biliary strictures: a prospective comparative study with bile and brush cytology. Am J Gastroenterol. 1996 Mar;91(3):465-7. PMID 8633492
- [Background] Tamada K, Tomiyama T, Wada S, Ohashi A, Satoh Y, Ido K, Sugano K. Endoscopic transpapillary bile duct biopsy with the combination of intraductal ultrasonography in the diagnosis of biliary strictures. Gut. 2002 Mar;50(3):326-31. doi: 10.1136/gut.50.3.326. PMID 11839709
- [Derived] Lenz P, Eckelskemper F, Erichsen T, Lankisch T, Dechene A, Lubritz G, Lenze F, Beyna T, Ullerich H, Schmedt A, Domagk D. Prospective observational multicenter study to define a diagnostic algorithm for biliary candidiasis. World J Gastroenterol. 2014 Sep 14;20(34):12260-8. doi: 10.3748/wjg.v20.i34.12260. PMID 25232260